CLINICAL TRIAL: NCT00027300
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Study to Determine the Safety and Efficacy of Natalizumab in Subjects With Relapsing-Remitting Multiple Sclerosis
Brief Title: Safety and Efficacy of Natalizumab in the Treatment of Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Elan Pharmaceuticals (Industry)
Responsible Party: Biogen Idec Medical Director, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-1801
Record Dates: First submitted 2001-11-30; First posted 2001-12-03 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Natalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Natalizumab 300 mg, IV
  Interventions: Drug: Natalizumab
- Group 2 (Placebo Comparator): Placebo IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Natalizumab — Natalizumab 300 mg IV infusion, every 4 weeks, for up to 116 weeks.
  Other Names: Tysabri
  Arms: Group 1
Drug: Placebo — Placebo, IV infusion, every 4 weeks, for up to 116 weeks.
  Arms: Group 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of natalizumab in the treatment of individuals who have been diagnosed with relapsing remitting multiple sclerosis (MS). It is hoped that natalizumab will prevent certain types of white blood cells from moving out of the bloodstream into organs, including the brain, that are being damaged by autoimmune disease (a disease in which the body's own immune system attacks certain organs). These white blood cells are thought to cause inflammation that can result in lesions (small areas of damage) in the brain. These lesions are thought to be the cause of relapses and disability in MS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS, as defined by McDonald et al., criteria # 1-4 (McDonald et al., 2001)
* Between the ages of 18 and 50, inclusive.
* Baseline EDSS score between 0.0 and 5.0, inclusive.
* Have experienced at least one relapse within the 12 months prior to randomization.
* Cranial MRI scan demonstrating lesion(s) consistent with MS.
* Have given written informed consent to participate in the study.

Exclusion Criteria:

* Primary progressive, secondary progressive, or progressive relapsing MS.
* MS relapse has occurred,in the opinion of the investigator, within 50 days prior to randomization and/or the subject has not stabilized from a previous relapse.
* A clinically significant infectious illness within 30 days prior to randomization.
* History of, or abnormal laboratory results indicative of any significant cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, gastrointestinal, dermatologic, psychiatric, renal and/or other major disease, that in the opinion of the investigator, would preclude the administration of a recombinant humanized antibody immunomodulating agent for 116 weeks.
* History of severe allergic or anaphylactic reactions or known drug hypersensitivity.
* Unable to perform the Timed 25-foot Walk, 9HPT, and PASAT 3.
* Abnormal blood tests performed at the Screening Visit.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 900 (Actual)
Dates: Start 2001-11; Primary Completion 2004-11 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
The primary objectives of this study are to determine whether natalizumab, when compared with placebo, is effective in reducing the rate of clinical relapses at 1 year and, in slowing the progression of disability at 2 years. | 1 year and 2 years

SECONDARY OUTCOMES:
Reduction in MRI changes and clinical relapses | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Panzara, MD, MPH, Study Director — Biogen; Chris Polman, MD, Principal Investigator — VU Medical Centre
Locations (53):
- United States (14):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - East Bay Region Associates in Neurology, Berkeley, California
  - UC Davis School of Medicine, Department of Neurology, Davis, California
  - Yale University School of Medicine, Department of Neurology, New Haven, Connecticut
  - University of Miami School of Medicine, Department of Neurology, Miami, Florida
  - University of Kansas Medical Center, Department of Neurology, Kansas City, Kansas
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Gimbel MS Center, Teaneck, New Jersey
  - CMRRC, Albuquerque, New Mexico
  - Oregon Health Sciences University, Department of Neurology, Portland, Oregon
  - Lehigh Valley Hospital, Neurosciences Research, Allentown, Pennsylvania
  - Texas Neurology, Dallas, Texas
  - University of Washington MS Research Center, Seattle, Washington
- Belgium (3):
  - Algemeen Ziekenhuis St. Jan, Bruges
  - LUC- University Centre, Diepenbeek
  - National MS Centrum, Melsbroek
- Canada (9):
  - Vancouver Hospital and Health Sciences Center UBC Pavilion, MS Clinical Research Group, Vancouver, British Columbia
  - Health Services Centre, Winnipeg, Manitoba
  - Kingston General Hospital, Neurology, Kingston, Ontario
  - University Hospital, London, Ontario
  - Sunnybrook and Women's College and Health Science Centre, Toronto, Ontario
  - University of Toronto, MS Clinic, St. Michael's Hospital, Toronto, Ontario
  - CHVO Hull Hospital, Québec, Quebec
  - MS Research Unit, Center for Clinical Research, Halifax
  - Family Medical Centre, Ottawa
- Czechia (9):
  - Faculty Hospital Brno Bohunice, Brno
  - Faculty Hospital St. Anne, Brno
  - Faculty Hospital of Hradec Kralove, Hradec Králové
  - Faculty Hospital Olomouc, Olomouc
  - Faculty Hospital Of Ostrava Poruba, Ostrava
  - Hospital Pardubice - Department of Neurology, Pardubice
  - Faculty Hospital Plzen - Clinic of Neurology, Pilsen
  - General Teaching Hospital - Neurological Department, Prague
  - Faculty Hospital Motol - Neurological Clinic, Prague
- France (2):
  - Hopital de la Timone, Service de Neurologie, Marseille
  - CHRU - Hopital de Pontchaillou, Service de Neurologie, Rennes
- Germany (2):
  - St. Josef-Hospital, Neurologische Klinik der Ruhruniversitat Bochum, Bochurn
  - Klinika Neurologii, Bydgoszcz
- Academisch Ziekenhuis VU, Amsterdam, Netherlands
- United Kingdom (13):
  - Institute of Neurology, Queen Square, London
  - The Royal London Hospital, Whitechapel, London
  - Atkin's Morely Hospital, Wimbledon, London
  - Oldchurch Hospital, Essex
  - Ipswich Hospital NHS Trust - Department of Clinical Neurology, Ipswich
  - St. James University Hospital, Department of Neurology, Leeds
  - Guy's Hospital, London
  - King's College Hospital, London
  - Kings College Hospital, Kings Neuroscience Center, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - The Radcliffe Infirmary, University Department of Clinical Neurology, Oxford
  - Royal Hallamshire Hospital, Sheffield
  - North Staffordshire Royal Infirmary - Neurology Department, Stoke-on-Trent

REFERENCES:
- [Background] Voloshyna N, Havrdova E, Hutchinson M, Nehrych T, You X, Belachew S, Hotermans C, Paes D. Natalizumab improves ambulation in relapsing-remitting multiple sclerosis: results from the prospective TIMER study and a retrospective analysis of AFFIRM. Eur J Neurol. 2015 Mar;22(3):570-7. doi: 10.1111/ene.12618. Epub 2014 Dec 15. PMID 25511792
- [Result] Polman CH, O'Connor PW, Havrdova E, Hutchinson M, Kappos L, Miller DH, Phillips JT, Lublin FD, Giovannoni G, Wajgt A, Toal M, Lynn F, Panzara MA, Sandrock AW; AFFIRM Investigators. A randomized, placebo-controlled trial of natalizumab for relapsing multiple sclerosis. N Engl J Med. 2006 Mar 2;354(9):899-910. doi: 10.1056/NEJMoa044397. PMID 16510744
- [Derived] Nakamura K, Sun Z, Hara-Cleaver C, Bodhinathan K, Avila RL. Natalizumab reduces loss of gray matter and thalamic volume in patients with relapsing-remitting multiple sclerosis: A post hoc analysis from the randomized, placebo-controlled AFFIRM trial. Mult Scler. 2024 May;30(6):687-695. doi: 10.1177/13524585241235055. Epub 2024 Mar 12. PMID 38469809
- [Derived] Strijbis EM, Coerver E, Mostert J, van Kempen ZLE, Killestein J, Comtois J, Repovic P, Bowen JD, Cutter G, Koch M. Association of age and inflammatory disease activity in the pivotal natalizumab clinical trials in relapsing-remitting multiple sclerosis. J Neurol Neurosurg Psychiatry. 2023 Oct;94(10):792-799. doi: 10.1136/jnnp-2022-330887. Epub 2023 May 12. PMID 37173129
- [Derived] Balcer LJ, Galetta SL, Polman CH, Eggenberger E, Calabresi PA, Zhang A, Scanlon JV, Hyde R. Low-contrast acuity measures visual improvement in phase 3 trial of natalizumab in relapsing MS. J Neurol Sci. 2012 Jul 15;318(1-2):119-24. doi: 10.1016/j.jns.2012.03.009. Epub 2012 Apr 21. PMID 22521274
- See also: The web site of the National Multiple Sclerosis Society, an organization dedicated to providing information to individuals with MS, their families and healthcare providers — http://www.nationalmssociety.org
- See also: MSActiveSource.com is a resource for news, information and disease management for all individuals touched by multiple sclerosis. This site is sponsored by Biogen. — http://www.msactivesource.com